CLINICAL TRIAL: NCT06479928
Title: The Mechanism of Interaction Between Arsenic Exposure and Gut Microbiota in Infants During Early Life
Brief Title: Interactions Between Environmental Exposures and Gut Microbiota in Early Life
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, xu xue, Vice Chief Physician, Peking University People's Hospital
Other Study IDs: PKUPH-X1
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Infant Development
Keywords: environmental exposure; gut microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — mother-infant stools, umbilical cord blood, placenta and hairs.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mother-infant cohorts (Cesarean section): Delivery mode, Cesarean section
  Interventions: Other: delivery mode
- Mother-infant cohorts (Natural delivery): Delivery mode, Natural delivery
  Interventions: Other: delivery mode

INTERVENTIONS:
Other: delivery mode — Based on delivery mode, we will divide them into two groups, including Cesarean section and Natural delivery.

SUMMARY:
Recruit the mothers and their infants who bron in Peking University People's Hospital from 2023 to 2026, to evaluate the interaction between environmental exposure and gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant woman

   * aged 20-40 years old
   * natural conception
   * single pregnancy
   * gestational age ≥36 weeks
2. Newborn

   * normal Apgar score
   * no serious congenital diseases

Exclusion Criteria:

-

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pregnant woman registered in Peking University People's Hospital will plan to give birth in the hospital.
Sampling Method: Probability Sample
Enrollment: 756 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Arsenic levels and Gut microbiota | Pregnancy (12, 24, 36 weeks) and infants (born, 1 week, and 1, 3, 6, 12, 24 months)
  Arsenic levels in biological samples; gut microbiota and metabolites in stools.

CONTACTS AND LOCATIONS:
Locations (1):
- The Peking University People's Hospital, Beijing, China